CLINICAL TRIAL: NCT06107465
Title: High Versus Low Dose Nitroglycerin in Management of Sympathetic Crashing Acute Pulmonary Edema
Brief Title: High Versus Low Dose Nitroglycerin in Acute Pulmonary Edema
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0108016
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Edema
Keywords: nitroglycein; dose; pulmonary edema
MeSH Terms: conditions — Pulmonary Edema | interventions — Nitroglycerin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose Nitroglycerin (Active Comparator): Initial dose of >100 mic/min will be initiated
  Interventions: Drug: Nitroglycerin
- Low dose Nitroglycerin (Active Comparator): Initial dose < 100 mic /min will be started
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — high dose Nitroglycerin

SUMMARY:
The goal of this randomized controlled trial is evaluate the out come of:

* Low dose (< 100 mic/min )versus
* High dose (> 100 mic/min) of nitroglycerin in management of patients with acute pulmonary edema presented to Emergency Department of Alexandria University Hospitals.

The main questions it aims to answer is:

* Time of resolution of high blood pressure, hypoxia, tacchypnea
* Need for invasive mechanical ventilation, ICU admission

DETAILED DESCRIPTION:
This single blind parallel randomized controlled trial will be conducted on (30 patients in each group) presented to Alexandria University Hospitals with acute pulmonary edema defined as: acute onset of dyspnea < 6 hrs, tacchypnea ( respiratory rate ≥30 breaths/min), bilaterak crepitations, O2 saturation < 90% on room air with associted sympathetic surge recognized by presence of tacchycardia, agitationa and blood pressure ≥ 160/90 mmHg

All patients included in the study will be allocated randomly using computer software with concealment of randomization in to two groups:

* Group (A): Low dose group Nitroglycerin at will be initiated at a rate <100 mic/min (15)
* Group (B): high dose group Initial dose > 100 mic /min (15) will be started Blood pressure will be measured for both groups every 15 minutes and dose adjusted accordingly, if the blood pressure starts to decrease continue infusion rate. In case of rising or constant blood pressure increase nitroglycerin by 20 mic/min every 15 min till blood pressure starts to decrease.

Initial, peak rate within the first hour, duration of IV nitroglycerin infusion will be recorded in both groups.

Initial and maximum dose of loop diuretic will be recorded in both groups.

Outcome:

Patients will be followed during ED stay to compare the two groups as regard:

* Time of resolution of high blood pressure.
* Resolution of hypoxia.
* Resolution of tachypnea.
* Need for invasive mechanical ventilation.
* Need for ICU admission.
* Length of hospital stay.
* Incidence of drug side effects as hypotension.
* Mortality.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (> 18 years) presented with sympathetic crashing acute pulmonary edema.

Exclusion Criteria:

1 - Patients indicated for emergency endotracheal intubation. 2-Patients with history of nitroglycerin allergy. 3-Preload dependent patients as patients with aortic stenosis. 4-Drug interaction with nitroglycerin as sildenafil, ergots. 5-Patients indicated for emergency percutaneous intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Resolution of symptoms | approximately 6 months
  ( hypoxia, high blood pressure and tacchypnea )

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrahman Hemeda, Resident, Principal Investigator — Alexandria University, Faculty of Medicine
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt